CLINICAL TRIAL: NCT05489796
Title: Comparison of Postoperative Side Effects and Analgesic Quality According to the Combination of Fentanyl and Ketorolac Versus Fentanyl After Laparoscopic Gynecologic Surgery
Brief Title: Bellomic PCA in Laparoscopic Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Principal Investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-2110-716-003
Record Dates: First submitted 2022-07-01; First posted 2022-08-05 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Laparoscopic Gynecological Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual group (Experimental): The two drugs are administered separately.
  Interventions: Drug: Fentanyl selector; Drug: Ketorolac continuous
- Single group (Active Comparator): One drug is administered alone.
  Interventions: Drug: Fentanyl selector; Drug: Fentanyl continuous

INTERVENTIONS:
Drug: Fentanyl selector — Selector (1 ml; Lock out 10 min): Fentanyl 200 mcg + N/S 16 ml = total 20 ml
Drug: Fentanyl continuous — Continuous (2 ml/hr): fentanyl 700 mcg + N/S 86 ml = total 100 ml
  Arms: Single group
Drug: Ketorolac continuous — Continuous (2 ml/hr): Ketorolac 180 mg + N/S 94 ml = total 100 ml
  Arms: Dual group

SUMMARY:
In laparoscopic gynecological surgery, when intravenous patient-controlled analgesia (IV-PCA) device is used after surgery, the degree of postoperative side effects and pain control is compared when a combination of fentanyl and ketorolac is administered compared to when fentanyl alone is used.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiology physical status 1 or 2
* Patients scheduled for gynecological laparoscopic surgery under general anesthesia
* Patients who applied for the use of IV-PCA after surgery

Exclusion Criteria:

* Patients with side effects of opioids
* Patients with hypersensitivity to aspirin or non-steroid anti-inflammatory drugs
* Patients with alcohol or drug dependence
* Patients with peptic ulcers, patients with gastrointestinal bleeding
* Patients with suspected cerebrovascular hemorrhage, organic disorders, or damage to the head related to increased intracranial pressure
* Symptoms of bronchial asthma or bronchospasm
* Patients with severe respiratory depression
* Moderate to severe renal impairment
* Patients with reduced blood volume or dehydration
* polyps in the nose
* angioedema
* Patients with or a history of the convulsive disease
* Patients for whom the use of neuromuscular blocking agents is contraindicated

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the occurrence of postoperative nausea | postoperative 0 hour, 2 hour, 6 hour, 12 hour, 24 hour
  Confirm the occurrence of postoperative nausea.
Change in the occurrence of postoperative vomiting | postoperative 0 hour, 2 hour, 6 hour, 12 hour, 24 hour
  Confirm the occurrence of postoperative vomiting.

SECONDARY OUTCOMES:
Change in the use of rescue antiemetics | postoperative 0 hour, 2 hour, 6 hour, 12 hour, 24 hour
  Investigate the use of rescue antiemetics.
Change of postoperative pain score | postoperative 0 hour, 2 hour, 6 hour, 12 hour, 24 hour
  Postoperative pain scores are scored on a scale of 0-10.
Change in the use of rescue analgesics | postoperative 0 hour, 2 hour, 6 hour, 12 hour, 24 hour
  Investigate the use of rescue analgesics.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea